CLINICAL TRIAL: NCT02302729
Title: Professor, Department of Pediatrics, University of Maryland School of Medicine
Brief Title: Early Child Development and Nutrition in Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Association for the Study and Prevention of HIV/AIDS (Other)
Responsible Party: Principal Investigator, Maureen Black, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00061322
Record Dates: First submitted 2014-10-31; First posted 2014-11-27 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Undernutrition
Keywords: Micronutrient intervention; Responsive feeding intervention; School readiness intervention
MeSH Terms: conditions — Malnutrition | interventions — Micronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Micronutrients No responsive feeding (Experimental): Micronutrient powder and no responsive feeding
  Interventions: Dietary Supplement: Micronutrients
- Placebo and Responsive Feeding (Placebo Comparator): Placebo (vitamin B2) and Responsive Feeding
  Interventions: Behavioral: Responsive feeding; Dietary Supplement: Placebo
- Micronutrients and Responsive caregiving (Experimental): Micronutrients and Responsive feeding intervention
  Interventions: Dietary Supplement: Micronutrients; Behavioral: Responsive feeding
- Placebo and No responsive caregiving (Placebo Comparator): Placebo and No responsive caregiving
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Micronutrients — Nutrient Quantity Nutrient Quantity Zinc 9 mg Copper 0.3 mg Iron 12.5 mg Vitamin D3 5 mg Folic Acid 160 mcg Vitamin E 5 mg Iodine 90 mcg Calcium 200 mg Vitamin A 250 mg Phosphorus 150 mg Vitamin C 40 mg Magnesium 40 mg Vitamin B12 0.9 mcg Selenium 17 mcg Thiamine 0.5 mg Manganese 0.17 mg Niacin 0.5 mg Biotin 8 mg Riboflavin 6 mg Vitamin B5 1.8 mg Vitamin B6 0.5 mg
  Arms: Micronutrients No responsive feeding; Micronutrients and Responsive caregiving
Behavioral: Responsive feeding — Strategy
  Mother ensures that feeding area is set up with infant and mother able to see one another.
  Mother mirrors the infant's facial expressions to attract the infant's attention.
  Mother interprets infant's behavior with a positive voice, "Oh, you like the spinach." Mother extends infant's behavior by saying, "Oh the cereal is all gone" and doing a consistent hand signal Mother models eating, makes positive comments in a nurturing tone. Mother offers finger food or use of utensil
  Arms: Micronutrients and Responsive caregiving; Placebo and Responsive Feeding
Dietary Supplement: Placebo — Riboflavin Vitamin B2
  Arms: Placebo and No responsive caregiving; Placebo and Responsive Feeding

SUMMARY:
Over 200 million children under the age of 5 years in low and middle-income countries do not reach their developmental potential, largely due to lack of adequate nutrients and lack of psychosocial stimulation. Stunting (length-for-age < -2 z-scores) is an indication of chronic undernutrition. Guatemala has the high rates of stunting in the Western Hemisphere (over 40%). This trial examines the effect of providing a micronutrient powder manufactured in Guatemala vs. placebo and an early learning environment vs. no early learning environment on the growth, health, and development of young children in Guatemala.

DETAILED DESCRIPTION:
The plan is to implement a clustered randomized placebo controlled trial with an infant phase (6-12 months of age) and a preschool phase (36-48 months of age). For the infant phase, the investigators will use ProPAN (Process for the Promotion of Child Feeding) in the development of the evaluation and intervention, with modifications as necessary for the Guatemalan context. ProPAN is a tool developed and distributed by the Pan American Health Organization to develop, implement, and evaluate interventions and programs to improve infant and young child diet and feeding. ProPAN includes four modules:

Module 1: Assessment Module 2: Testing Recipes and Recommendations Module 3: Intervention Module 4: Monitoring and Evaluation

For the preschool phase, the investigators will use an evidence-based school readiness intervention (Little By Little) that has been shown to be effective with Hispanic preschoolers. The intervention will be implemented through the Association for the Prevention and Study of HIV/AIDS who will train and supervise the community health workers. By working directly with a local non-profit organization, the project will be well positioned to inform strategies to scale up the intervention on a community wide basis, if beneficial effects are shown.

The project examines the effects of an integrated intervention that includes both micronutrient powder added to food and responsive feeding for infants or school readiness for preschoolers. The primary aim is to examine how an integrated micronutrients + responsive feeding/school readiness intervention changes the development (primary outcome), growth and micronutrient status (secondary outcomes) of young children. The investigators will focus on infants (6-12 months) when the risk for micronutrient deficiencies is high, as they transition from breast feeding to complementary feeding and the family diet. The investigators will focus on preschoolers (36-48 months) to examine if micronutrients + a school readiness intervention can improve children's school readiness skills. The design includes neighborhood clusters randomized into four groups: 1) micronutrients plus responsive feeding/school readiness 2) micronutrients only, 3) placebo plus responsive feeding/school readiness, and 4) placebo only.

The investigators will test the following hypotheses:

1. Children in the two micronutrients groups have better change from baseline in development (primary outcome), growth and micronutrient status (secondary oitcomes), than children in the two placebo groups.
2. Mothers and children in the two responsive feeding/school readiness groups have better change from baseline measures of child development than those in the two control groups.
3. The impact of the responsive feeding/school readiness intervention is greater in the micronutrient groups than in the placebo groups. Children in the micronutrients plus responsive feeding/school readiness group have better change from baseline in development than children in any of the other three groups.

ELIGIBILITY:
Inclusion Criteria:

* Child speaks Spanish.
* Child is age 6-12 months or age 36-48 months.
* Child must be undernourished (length and height for age < -1 z-score).
* Child does not have any obvious health or developmental problems that would interfere with growth, nutrition, or development.
* Child will remain in the area for the subsequent year.
* Parent or legal guardian of the child is age 18 years or older.
* Parent or legal guardian speaks and understands Spanish.
* Parent or legal guardian lives with child in study community.

Exclusion Criteria:

* Child is not age 6-12 months or 36-48 months.
* Child has severe stunting (length and height for age < -3 z-scores).
* Child has identified conditions that could interfere with their development and growth.
* Child is severely anemic (hemoglobin < 7).

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1730 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2015-12-08 (Actual); Study Completion 2015-12-08 (Actual)

PRIMARY OUTCOMES:
Change in cognitive, motor, social-emotional development from baseline to 12 months | Baseline, 12 months
  Cognitive and social-emotional assessments

SECONDARY OUTCOMES:
Change in Growth from baseline to 12 months | Baseline, 12 months
  Weight, length/height
Change in micronutrient status from baseline to 12 months | Baseline, 12 months
  Blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Maureen M Black, Ph.D., Principal Investigator — Uniersity of Maryland, Baltimore
Locations (1):
- APEVIHS (Association for the Prevention and Study of HIV/AIDS), Retalhuleu, Guatemala

REFERENCES:
- [Background] Unable to connect to PubMed to validate , last attempt on November 19, 2014 at 3:47 PM EST